CLINICAL TRIAL: NCT03538418
Title: Enhancing the Physical Activity Levels of Community-dwelling Older People With Frailty Through an Exercise Intervention With or Without a Wearable Activity Tracker (WAT)-Based Intervention: a Feasibility and Pilot Study
Brief Title: Enhancing Physical Activity Levels of Frail Older People With a Wearable Activity Tracker-based Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSEARS20180320006
Record Dates: First submitted 2018-04-19; First posted 2018-05-29 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Frail Elderly
Keywords: Frailty; Wearable technology; Physical activity; Behaviour change
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: A two-arm parallel (single-blinded) cluster randomized controlled trial involves two groups of participants (the WAT group and the control group). Six community centres, which provide similar types of community care and social support services for community-dwelling older people, will be invited by a convenience method to work as collaborators in this study. Using computer-generated random numbers, a biostatistician not affiliated with this study will randomize the centres into either: the control or the experimental groups. Therefore, duing the trial, participants in one group receive intervention "in parallel" to participants in the other group (control group).
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is blinded to the group allocations will assess the participants' outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WAT group (Experimental): The WAT group will receive a 3-month WAT-based exercise training programme, which includes 12 weekly exercise training sessions (an hour each) in addition to 2 face-to-face sessions followed by weekly to monthly telephone sessions offering support on dealing with technical issues and BCTs (7 session in total). The WAT group will be left to use the WAT on their own for 3 months during the follow-up period.
  Interventions: Other: WAT
- Control group (No Intervention): The control group will receive a 3-month exercise training programme without a WAT, which also includes 12 weekly exercise training sessions (an hour each) in addition to 7 face-to-face and telephone sessions offering support for BCTs.

INTERVENTIONS:
Other: WAT — The WAT intervention consists of 12 weekly WAT-based exercise sessions and 7 sessions of support for BCTs and technical issues.
  Arms: WAT group

SUMMARY:
This study aims to investigate the feasibility, acceptability, and preliminary effects of a Wearable Activity Tracker (WAT)-based exercise intervention to increase physical activity levels in frail or pre-frail older people. One group of participants will receive a WAT-based exercise intervention incorporated with the support of behavioral change techniques (BCTs) and technical issues, while the other group will receive only an exercise intervention incorporated with BCTs support.

DETAILED DESCRIPTION:
Six community centres, which provide similar types of community care and social support services for community-dwelling older people, will be invited by a convenience method to work as collaborators in this study. Using computer-generated random numbers, a biostatistician not affiliated with this study will randomize the centres in a 1:1 ratio into either: the control or the experimental groups (WAT group).

The WAT group will receive a 3-month exercise programme plus WAT intervention which aims to strengthen the participants' motivation to develop the intention to gradually increase their physical activity levels to eventually meet the level recommended for older people by the American Heart Association (AHA). Two face-to-face sessions followed by weekly to monthly telephone sessions offering support on dealing with technical issues and BCTs will be arranged for the experimental group. The additional technical support given alongside the WAT intervention will be gradually withdrawn from the participants. Eventually, all additional measures to support the use of WATs among participants will be stopped. Participants will be left to use the WAT on their own for 3 months during the follow-up period. In addition, they will receive a weekly 45-60 minute center-based structured exercise programme for 3 months, which is designed according to the AHA's recommendations on exercise for older people.

The control group will receive another 3-month exercise programme with face-to-face, and telephone-delivered BCTs follow-up sessions, with the number and timing of all sessions similar to that in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older people aged > 65 years;
* able to communicate in Cantonese to ensure that they understand our instructions;
* able to walk with or without an assistive device and able to complete the Time Up and Go (TUG) test with no specific cutoff point to ensure that their mobility and balance is good enough to join the exercise training;
* able to use a smartphone;
* with daily walking steps less than 7000, and
* in a pre-frail or frail state as determined using the Fried Frailty Index; including: i) having experienced an unintentional loss of 10% of body weight in the past year; ii) exhaustion: by answering 'Yes' to either 'I felt that everything I did was an effort', or 'I could not get going in the last week'; iii) a slow walk time: with an average walking speed in the lowest quintile stratified by median body height; iv) reduced grip strength: with maximal grip strength in the lowest quintile stratified by the body mass index quartile; and v) a Physical Activity Scale for Elderly-Chinese (PASE-C) score in the lowest quartile (i.e., < 30 for men and < 27.7 for women). The presence of 1-2 indicates pre-frailty, > 3 items indicates frailty.

Exclusion Criteria are older people who:

* have any physical conditions that hamper their performance of the exercise programme or use of the WAT, such as visual or hearing problems.
* regularly engage in moderately intense exercise (such as hiking, Tai Chi) for > 3 hours per week.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of using the activity tracker | Throughout the 3-month programme
  The number of days that a participant in the experimental group wears and syncs the device divided by the number of intervention days.
Recruitment rate | Enrollment date
  The proportion of participants who consent to join the study over the eligible participants.
Attrition rate | At the end of the 3-month programme
  The percentage of participants who withdraw from the study and their reasons for withdrawing.
Adherence to the exercise regimen | Throughout the 3-month programme
  Exercise adherence will be assessed by the training session attendance, the participants' adherence to the desired levels of MVAP as suggested by the physical trainer and the exercise diary.
Occurrence of adverse events at home | Throughout the 3-month programme
  Any adverse events at home will be recorded.
Change of activity levels (total steps) measured by ActiGraph wGT3X accelerometer. | Change from Baseline Activity Level at 1 week, *1 month and * 3 month post-intervention (* only for the experimental group)
  The participants' total steps will be collected.
Change of activity levels (activity) measured by ActiGraph wGT3X accelerometer. | Change from Baseline Activity Level at 1 week, *1 month and *3 month post-intervention(* only for the experimental group)
  The time spent in activities of different intensity (sedentary, light, moderate and vigorous) will be collected.
Change of sleep quality (sleep time) measured by ActiGraph wGT3X accelerometer. | Change from Baseline Activity Level at 1 week, *1 month and *3 month post-intervention. (* only for the experimental group)
  The participant's total sleep time will be collected.
Change of sleep quality (wake after sleep onset) measured by ActiGraph wGT3X accelerometer. | Change from Baseline Activity Level at 1 week, *1 month and *3 month post-intervention.(* only for the experimental group)
  The frequency of wake after sleep onset of the participant will be collected.

SECONDARY OUTCOMES:
Activity levels (total steps) assessed by activity monitor (Fitbit) | Throughout the 3-month programme
  The total steps per week of an individual will be collected.
Activity levels (total walking distance) assessed by activity monitor (Fitbit) | Throughout the 3-month programme
  The total walking distance per week of an individual will be collected.
Activity levels (time spent in different heart rate zones) assessed by activity monitor (Fitbit) | Throughout the 3-month programme
  The time spent in different heart rate zones of an individual will be collected.
Participants' lower-limb strength will be assessed using the 30-second chair stand test | Baseline, at 1 week, *1 month and* 3 month post-intervention (* only for the experimental group)
  Participants will be asked to stand up and sit down as many as they can within 30 seconds on a standard chair. The total number of standing up from a chair will be counted. More number indicates better lower-limb strength
Participants' upper-limb strength will be assessed using a handheld Jamar Hydraulic Hand Dynamometer | Baseline, at 1 week, *1 month and *3 month post-intervention (* only for the experimental group)
  It will be measured by handheld Jamar Hydraulic Hand Dynamometer with kilogram (kg). Greater force in kg indicates better upper-limb strength
Participants' functional mobility will be measured by the timed-up-and-go-test | Baseline, at 1 week, *1 month and *3 month post-intervention
  Record the time in second that participants complete the timed up and go test to indicate their functional mobility
Participants' gait speed will be measured by the 2 minutes walk test | Baseline, at 1 week, 1 month and 3 month post-intervention (* only for the experimental group)
  Record the time in second that participants complete the 2 minutes walk test to indicate the their gait speed.
Participants' exercise self-efficacy will be measured using Chinese Self-Efficacy for Exercise (CSEE) scale | Baseline, at 1 week, *1 month and *3 month post-intervention (* only for the experimental group)
  The CSEE scale contains of 9 items. Each item is rated on 11-point Liker scale from 0 = no confidence to 10 = full of confidence. All item scores are summed to get the total score which ranges from 0 to 90 with a higher score indicates higher exercise self-efficacy
Participants' frailty level will be assessed using Fried Frailty Index (FFI) | Baseline, at 1 week, *1 month and *3 month post-intervention (* only for the experimental group)
  Fried Frailty Index includes: i) an unintentional loss of 10% of body weight in the past year; ii) exhaustion: by answering 'Yes' to either 'I felt that everything I did was an effort', or 'I could not get going in the last week'; iii) a slow walk time: with an average walking speed in the lowest quintile stratified by median body height; iv) reduced handgrip strength: with maximal grip strength in the lowest quintile stratified by body mass index quartile; and v) the Physical Activity Scale for the Elderly-Chinese (PASE-C) score in the lowest quintile (i.e., < 30 for men and < 27.7 for women).
Participants' self-reported sedentary behavioral and physical activity will be assessed using Global Physical Activity Questionnaire-Chinese version (C-GPAQ) | Baseline, at 1 week, *1 month and *3 month post-intervention (* only for the experimental group)
  The C-PAQ comprises 16 questions designed to estimate an individual's self-perceived level of physical activity in three domains (occupational, transport-related and discretionary or leisure time).
Participants' motivation to engage in physical activity using of the Behavioral Regulation in Exercise Questionnaire-2 (C-BREQ-2) | Baseline, at 1 week, *1 month and *3 month post-intervention (* only for the experimental group)
  C-BREQ-2 is a 19-item questionnaire assessing five dimensions: amotivation, external regulation, introjected regulation, identified regulation, and intrinsic regulation. Each item is rated on a 5-point scale ranging from 0 = "not true for me" to 4 = "very true for me", with higher scores indicative of higher motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Justina LIU, Dr., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic Universtiy, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Informed Consent Form (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03538418/ICF_000.pdf
  • Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03538418/SAP_001.pdf
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03538418/Prot_002.pdf